CLINICAL TRIAL: NCT04315402
Title: The Impact of Provider Demographics on Patients' Continuity of Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 19-105
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Race Concordant Patient-provider Relationship; Race Discordant Patient-provider Relationship; Rate of No-show at Follow-up Visits
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (provider-patient concordant)
  Interventions: Other: prospective, descriptive study via survey
- Group 2 (provider-patient discordant)
  Interventions: Other: prospective, descriptive study via survey

INTERVENTIONS:
Other: prospective, descriptive study via survey — * Survey administered at check out.
  * Patient's rate of follow-up data gathered via chart review.

SUMMARY:
The race concordance of providers to their patients impacts a patient's investment and agency in the patient-provider relationship. The mistrust of medicine within the African American population remains and patients feel unengaged in their care. Race concordant provider-patient rela-tionships would improve the equity of patient care in our clinic.

DETAILED DESCRIPTION:
The patients of the obstetrics and gynecology resident clinic at Good Samaritan Hospital have a poor follow-up rate for their gynecologic and prenatal care visits. In addition, patients oftentimes voice frustration over the care that they receive and sometimes remark that they feel their provider was "racist." These patients often have complex social situations that cannot be solved in one office visit but perhaps the providers' ability to gain the trust of the minority patients is inadequate. The residents in the OB/GYN program are 80% white with no African American representation. If patients are unable to connect with caregivers due to cross-cultural differences, this could be remedied by training current residents in cross-cultural communication or re-cruitment of a resident class more representative of the majority African American patient population. This project will provide perspective on the minority patients' needs in the provider-patient relationship and allow providers to reexamine their ability to gain trust with the ultimate goal to increase follow-up rates. Follow-up rates for prenatal care are directly linked to improved maternal and fetal outcomes. The investigators goals are threefold: to gain clarity on whether or not a more diverse resident group would be helpful in gaining the trust of patients, to assess the current state of the well-established historical and generational mistrust of medical care by the African American patients of the clinic, and to explore how patient perception of their provider impacts their rate of follow up in the large community hospital clinic.

ELIGIBILITY:
Inclusion criteria

* Female Patient seeing OB/GYN resident at FMC
* 18 years or older
* <36 weeks pregnant or GYN patient
* If GYN patient, must have problem requiring follow-up within 6 months
* Have not previously completed the survey

Exclusion criteria

* Less than 18 years of age
* High risk clinic patients (Tuesday afternoons)
* Patients without a follow-up less than 6 months as scheduled at check out

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients of the Faculty Medical Center seeing OB/GYN residents
  * Those requiring follow-up (less than 6 months)
Sampling Method: Probability Sample
Enrollment: 415 (Estimated)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Patient's rate of follow-up | 6 months
  Whether or not patient was present at their next scheduled GYN or OB follow-up appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Nima Patel, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No